CLINICAL TRIAL: NCT03950427
Title: PARQuit Smoking Cessation Intervention for Adults With Serious Mental Illness
Acronym: PARQuit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T29IP0235; 22637 (Other: University of California, San Francisco); NCI-2022-02281 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation; Smoking, Tobacco; Mental Illness; Tobacco Use Disorder
Keywords: smoking cessation; serious mental illness
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking; Mental Disorders; Tobacco Use Disorder | interventions — Bupropion; Counseling

STUDY DESIGN:
Intervention Model Description: This study is a pilot, randomized controlled trial (RCT) to examine the feasibility and potential efficacy of an application of a videogame-based group physical activity intervention for smoking cessation in adults with SMI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Game-based Physical Activity Group (Active Comparator): The game-based physical activity group, will play active games using the Kinect for Xbox 360 game system or outdoors in a public park. Each game group will be facilitated by the study coordinator, the principal investigator or other study staff.
  Participants in this group will also receive bupropion and counseling for smoking cessation.
  Interventions: Behavioral: Videogame-based physical activity; Drug: Bupropion; Behavioral: Counseling
- Sedentary Videogame Group (Placebo Comparator): The sedentary videogame group will play games while seated using the Xbox 360 game system (without the Kinect sensor) or seated outdoors in a public park. Each sedentary videogame group will be facilitated by study staff.
  Participants in this group will also receive bupropion and counseling for smoking cessation.
  Interventions: Behavioral: Sedentary videogame; Drug: Bupropion; Behavioral: Counseling

INTERVENTIONS:
Behavioral: Videogame-based physical activity — videogame-based physical activity
  Arms: Game-based Physical Activity Group
Behavioral: Sedentary videogame — sedentary videogame
  Arms: Sedentary Videogame Group
Drug: Bupropion — Bupropion
  Other Names: Wellbutrin; Zyban
Behavioral: Counseling — Counseling for smoking cessation

SUMMARY:
This is a research study about a smoking cessation program tailored for adults with serious mental illness (SMI). The program uses a Videogame-based Physical (VIP) activity, smoking cessation counseling, and medication (bupropion),

DETAILED DESCRIPTION:
The purpose of this study is to learn more about how adults with serious mental illness respond to a smoking cessation program combining a game-based Physical activity, counseling for smoking cessation, and a medication (bupropion or NRT) for smoking cessation.

Study participants will receive counseling to quit smoking and a medication to help decrease cravings and withdrawal. Additionally, participants will be randomly selected to participate in either a game-based physical activity group or a game group where the participants sit to play the games.

Participants will be in this study for 12 weeks total. There are 3 assessment visits (2 hours each) at the beginning of the study, 6 weeks after starting, and at the end of the 12 weeks. There will be 8 30- minute counseling sessions during the 12 weeks. The hour-long videogame groups will be held 3 times a week for 12 weeks (36 sessions). Upon completion of the 12-week program, there will be a 1-2 hour group interview. The total time commitment is 48 hours over the course of the 12-week study.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of a Serious Mental Illness (SMI)*
* 18 years and older
* Smoking at least five cigarettes per day for the past 6 months
* Willingness to set a quit date
* Not currently taking bupropion or using nicotine replacement therapy (NRT)
* Current participant in the residential or day treatment program at a Progress Foundation program with the intention to continue in the residential or day treatment program for at least the 12 week intervention period
* Capacity to consent.

  * SMI is characterized by the American Psychological Association as distinct conditions that require routine management, produce functional impairment, and interfere with quality of life. Individuals that typically meet the criteria of SMI have illnesses that include schizophrenia, schizoaffective disorder, psychotic disorders, major depressive disorders, bipolar disorders, and borderline personality disorder.

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Diagnosis of seizure disorder, history of anorexia/bulimia, undergoing abrupt discontinuation of ethanol or sedatives, other conditions that increase seizure risk (e.g., arteriovenous malformation (AVM), severe head injury, central nervous system (CNS) tumor)
* use of Monoamine oxidase (MAO) inhibitors (concurrently or within 14 days of discontinuing either bupropion or the MAO inhibitor)
* Planning to become pregnant during the study period
* Previous participation in the videogame-based physical activity intervention.
* Known medical conditions or other physical problems that need special attention in an exercise program (e.g. prior myocardial infarction, uncontrolled hypertension, history of angioplasty, history of angina, use of nitroglycerin to treat angina)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Total number of videogame sessions attended | Up to 12 weeks
  Feasibility will be measured with a total count of sessions attended. The graduate student researcher (GSR) will document participant attendance.
Total minutes of videogame sessions attended | Up to 12 weeks
  Feasibility will be measured with a sum of minutes attended. The GSR will monitor and document the times when participants enter and leave the sessions.
Week-6 Self-report acceptability rankings of the videogames | 6 weeks
  This internally developed acceptability questionnaire has 7 questions. Three questions use a 1 to 5 scale with 1 indicating least acceptable and 5 indicating most acceptable, for a possible total range of 3-15. The remaining open-ended questions are scored using qualitative thematic analysis.
Week-12 Self-report acceptability rankings of the videogames | 12 weeks
  This internally developed acceptability questionnaire has 7 questions. Three questions use a 1 to 5 scale with 1 indicating least acceptable and 5 indicating most acceptable, for a possible total range of 3-15. The remaining open-ended questions are scored using qualitative thematic analysis. Used to measure change from week-6 to week-12.
Week-6 Tobacco reduction and abstinence | 6 weeks
  The investigators will ask about the number of cigarettes, even a puff, smoked in the past week (7-day abstinence) or use of any form of tobacco or alternative tobacco product e.g., e-cigarette or heat not burn. Salivary cotinine levels will be measured to determine abstinence from smoking.
Week-12 Tobacco reduction and abstinence | 12 weeks
  The investigators will ask about the number of cigarettes, even a puff, smoked in the past week (7-day abstinence) or use of any form of tobacco or alternative tobacco product e.g., e-cigarette or heat not burn. Salivary cotinine levels will be measured to determine abstinence from smoking.
Mean Scores at Baseline on the Brief Psychiatric Rating Scale (BPRS) | Baseline interview with the participant and observations of the participant's behavior over the previous 2-3 days.
  The Semi-Structured Interview for Brief Psychiatric Rating Scale is completed by the PI or trained research staff and assesses the number and severity of psychiatric symptoms. It consists of 24 items that are rated from 1 (not present) to 7 (extremely severe), and the items are summed for a total psychopathology score, with a possible range from 24-168 and a higher score indicating a higher severity of illness.
Mean scores at Week-6 on the Brief Psychiatric Rating Scale (BPRS) | 6 weeks
  The Semi-Structured Interview for Brief Psychiatric Rating Scale is completed by the PI or trained research staff and assesses the number and severity of psychiatric symptoms. It consists of 24 items that are rated from 1 (not present) to 7 (extremely severe), and the items are summed for a total psychopathology score, with a possible range from 24-168 and a higher score indicating a higher severity of illness.
Mean scores at Week-612 on the Brief Psychiatric Rating Scale (BPRS) | 12 weeks
  The Semi-Structured Interview for Brief Psychiatric Rating Scale is completed by the PI or trained research staff and assesses the number and severity of psychiatric symptoms. It consists of 24 items that are rated from 1 (not present) to 7 (extremely severe), and the items are summed for a total psychopathology score, with a possible range from 24-168 and a higher score indicating a higher severity of illness.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Leutwyler, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No